CLINICAL TRIAL: NCT04694001
Title: Evaluation of the Use of the Atalante Exoskeleton in Patients Presenting an Hemiplegia Due to Cerebrovascular Accident
Acronym: INSPIRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wandercraft (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: INSPIRE
Record Dates: First submitted 2020-12-28; First posted 2021-01-05 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Stroke; Stroke, Acute; Stroke, Subacute; Chronic Stroke
Keywords: Robotics; Rehabilitation; Physiotherapy; Powered exoskeleton; Walking; Exercises; Ambulation; Stroke; Acute stroke; Subacute stroke; Chronic stroke
MeSH Terms: conditions — Stroke; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hemiplegia due to Cerebrovascular Accident (CVA) (Other)
  Interventions: Device: Use of the Atalante exoskeleton

INTERVENTIONS:
Device: Use of the Atalante exoskeleton — A session includes stand-up, walks, exercises with or without the assistance of the exoskeleton, rotation, side and back step, squat and sitting.

SUMMARY:
The INSPIRE study is interventional, European, prospective, open, multicentric, each patient being his/her own control.

It is conducted to assess the safety and performance of the Atalante exoskeleton system in patients presenting an hemiplegia due to cerebrovascular accident. The primary endpoint is defined by the reported adverse events.

The study will include 40 patients and takes place in six rehabilitation centers (4 in France, 1 in Luxembourg, 1 in Belgium).

ELIGIBILITY:
Inclusion Criteria:

* Patient with hemiplegia due to cerebrovascular accident, occurred two weeks ago or more, follow up in a rehabilitation center or in a hospital (inpatient or outpatient),
* Patient presenting a FAC score of 0, 1, 2 or 3,
* Patient whose etiological evaluation of the stroke has been complete,
* Adult patient ≥18 years old,
* Patient able to read and write in at least one of the languages of the country and who have signed an informed consent form.

Exclusion Criteria:

* Individuals with severe spasticity of adductor muscles, hamstring, quadriceps and triceps surae. Severe spasticity is defined by a score greater than 3 on the modified Ashworth scale,
* Pregnant women
* Individuals with history of osteoporotic fracture and pathology or treatment causing secondary osteoporosis,
* Pressure Ulcer of Grade I or higher according to the National Pressure Ulcer Advisory Panel (NPUAP) International Pressure Ulcer Classification System- European Pressure Ulcer Advisory Panel (EPUAP), in areas of contact with the Atalante system,
* Severe aphasia limiting ability to express needs or to fulfil questionnaires, at the discretion of the physician.
* Patient with a cardiac or respiratory contraindication to physical exertion,
* Patient with a score below 18 on the Mini Mental State test,
* Patient unable to deliver his/her consent,
* Patient under legal protection,
* Patient participating at the same time in another study,
* Patients with morphological contraindications to the use of the Atalante exoskeleton.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2022-03-28 (Actual); Study Completion 2022-03-28 (Actual)

PRIMARY OUTCOMES:
The primary objective is to evaluate the incidence of treatment-emergent adverse events. | Throughout study completion, an average of 6 days
  The primary endpoint is measured through reported Adverse Events (AEs) including adverse events (AEs), adverse device effects (ADEs), serious adverse events (SAEs), serious adverse device effects (SADEs), adverse procedure effects (APE), and new findings (NFs).

SECONDARY OUTCOMES:
Evaluate the patient's ability to walk without the Atalante exoskeleton | At study start, day 1 and at study completion, up to 6 days
  Evaluation of the walk performance with the Functional Ambulation Category (FAC) at baseline and session 6 (from 0 to 5, 0 being "patient cannot walk" and 5 "patient can walk independently anywhere")
Evaluate the patient's gait speed without the Atalante exoskeleton | At study start, day 1 and at study completion, up to 6 days
  Evaluation of the gait speed measured without the Atalante exoskeleton in 10-Meter Walk Test (10MWT) at baseline and session 6
Evaluate the patient's endurance without the Atalante exoskeleton | At study start, day 1 and at study completion, up to 6 days
  Evaluation of the covered distance without the Atalante exoskeleton measured in 6-Minute Walk Test (6MWT) at baseline and session 6
Evaluate the patient's static and dynamic balance without the Atalante exoskeleton | At study start, day 1 and at study completion, up to 6 days
  Evaluation of static and dynamic balance without the Atalante exoskeleton measured with the Berg Balance Scale (BBS) at baseline and session 6 (0-20 on the BBS represents balance impairment; 21-40 on the BBS represents acceptable balance; 41-56 on the BBS represents good balance)
Evaluate the patient's spasticity | At study start, day 1 and at study completion, up to 6 days
  Evaluation of the spasticity of the adductor muscles, hamstrings, quadriceps, and triceps surae measured with Modified Ashworth Scale at baseline and session 6
  0 No increase in muscle tone
  1. Slight increase in muscle tone, manifested by a catch and release or by minimal resistance at the end of the range of motion (ROM) when the affected part(s) is moved in flexion or extension 1+ Slight increase in muscle tone, manifested by a catch, followed by minimal resistance throughout the remainder (less than half) of the ROM
  2. More marked increase in muscle tone through most of the ROM, but affected part(s) easily moved
  3. Considerable increase in muscle tone, passive movement difficult
  4. Affected part(s) rigid in flexion or extension
Evaluate the patient's pain | At study start, day 2 and at study completion, up to 6 days
  Evaluation of the pain measured before and after sessions 1 to 5 using the Visual Analogical Scale-Pain.
  The patient is asked to make pain ratings between "No Pain" and "Maximum pain imaginable", , with "No pain" corresponding on 0 on the caregiver side and and "Maximum pain imaginable" to 10 on caregiver side.
Evaluate the patient's capability to stop the exoskeleton on time using the remote | At study mid term, up to 5 days
  Evaluation of the patient's capability to stop the exoskeleton, on time using the remote at session 5
Evaluate the patient's satisfaction and perceptions upon completion of a locomotor training program with the Atalante exoskeleton | At study completion, up to 6 days
  Evaluation of the satisfaction et perceptions via a questionnaire specific to the use of robotics exoskeleton at session 6.
  Questions are answered on a 7-level Likert scale.
Evaluate the use of the Atalante exoskeleton | At study start, day 2 and at study completion, up to 6 days
  Collection of data relating to the patient's walking parameters and level of assistance with the Atalante exoskeleton during sessions 1 to 5
Evaluate the patient's skin condition to monitore the pressure points the patient may have with the contact of the exoskeleton. | At study start, day 2 and at study completion, up to 6 days
  The operator will perform a visual monitoring of the patient's skin to identify potential cutaneous morbidity at pressure points the patient may have with the exoskeleton before and after sessions 1 to 5.
Evaluate the patient's level of anxiety and depression | At study start, day 1 and at one week afetr the study completion, up to 12 days
  Assessment of patient anxiety and depression by means of the Hospital Anxiety and Depression (HAD) scale at baseline and one week after the 5th session

CONTACTS AND LOCATIONS:
Locations (6):
- Cliniques universitaires Saint-Luc, Brussels, Belgium
- France (4):
  - Centre Jacques Calvé - Fondation Hopale, Berck
  - Centre de Médecine Physique et de Réadaptation, Pionsat
  - Centre mutualiste de Rééducation et de Réadaptation de Kerpape, Ploemeur
  - Hôpital La Musse, La Renaissance Sanitaire, Saint-Sébastien-de-Morsent
- Rehazenter, Luxembourg, Luxembourg

REFERENCES:
- [Derived] Lejeune T, Nuic D, Dehem S, Previnaire JG, Cuenot C, Debugne T, Kaps J, Paul B, Pean V, Perez SS, Juhel F, Tatsidou S, Kerdraon J. Hands-free Atalante exoskeleton in post-stroke gait and balance rehabilitation: a safety study. J Neuroeng Rehabil. 2025 Apr 12;22(1):82. doi: 10.1186/s12984-025-01621-z. PMID 40221748